CLINICAL TRIAL: NCT04823728
Title: Immunogenetic Characteristics in Autoimmune Encephalitis and Related Disorders: HLA Analysis: Part II
Brief Title: HLA Analysis in Autoimmune Encephalitis and Related Disorders: Part II
Acronym: ICARE-II
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0826
Record Dates: First submitted 2021-03-26; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Autoimmune Encephalitis; Paraneoplastic Neurological Syndrome
Keywords: Autoimmune encephalitis; Paraneoplastic neurological syndromes
MeSH Terms: conditions — Autoimmune Diseases of the Nervous System

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood collected at diagnosis time
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Autoimmune encephalitis and paraneoplastic neurological syndromes: Patients with well-characterized antibodies against onconeural antigens, synaptic or cell-surface antigens
  Interventions: Genetic: Autoimmune encephalitis and paraneoplastic neurological syndromes

INTERVENTIONS:
Genetic: Autoimmune encephalitis and paraneoplastic neurological syndromes — This is a non-interventional study involving biological samples (DNA). Samples are already stored in biobank repositories and collected as part of "good clinical practice" in the diagnostic process of patients with suspected autoimmune encephalitis, meaning that the standard diagnostic and therapeutic approaches will not be altered in the selected study population. Patients have already gave explicit written consent for biological specimens sampling and storage at the "Centre de Ressources Biologiques des Hospices Civils de Lyon" (CRB-HCL)/NeuroBioTec (including tissue, cells or biological fluids) and genetic analysis for research purposes (e.g. involving genes related to the disease for which the patient was followed). Additionally, patients will be informed about the present study.

SUMMARY:
Autoimmune encephalitis (AE) are characterized by subacute onset of memory deficits, altered mental status or psychiatric symptoms, frequently associated with seizures, inflammatory cerebrospinal fluid and in cases with prominent limbic involvement, typical magnetic resonance imaging. Several autoantibodies (Abs) may be detected in AE, although its detection is not mandatory to establish a diagnosis. These Abs mainly recognize different synaptic and cell-surface proteins in the central nervous system, and are thought to be pathogenic as they alter the normal location or function of its antigens. Paraneoplastic neurological syndromes (PNS) are immune-mediated, remote complications of cancer. The clinical presentation is highly diverse, from central nervous system disorders (limbic encephalitis, cerebellar ataxia) to peripheral neuropathies and neuromuscular junction diseases. Two different kinds of Abs are associated with PNS: a first group known as onconeural Abs, which recognize intracellular antigens and are thought not to be pathogenic; and a second one whose targeted synaptic and cell-surface antigens shared with some non-paraneoplastic AE.

The primary trigger of the immune response is unknown for most of AE. In addition to acquired susceptibility such as herpes simplex encephalitis, genetic predisposition may also be important in the pathogenesis of AE. Human leukocyte antigen (HLA) is the genetic factor most frequently associated with autoimmune diseases, due to its genetic complexity and key role in the adaptive immune response. Others and we already described the HLA haplotypes associated with three types different of AE: anti-leucine-rich glioma inactivated 1 (LGI1), anti-contactin-associated protein-like 2 (CASPR2), and anti-glutamic acid decarboxylase (GAD). Nevertheless, the genetic predisposition of many other AE has not been investigated yet.

Cancer is considered as the trigger of the immune response that lead to PNS development, as the neural antigens recognized by the onconeural Abs are also expressed by tumor cells. Nevertheless, it is still unknown why some patients develop PNS and others do not, even if they present the same histological type of tumor, suggesting that some particular, maybe genetic, characteristics of the patients may play a role in this susceptibility. Furthermore, there is already evidence that, for those neurological diseases that may appear either as PNS or as non-paraneoplastic autoimmune disorder (i.e. Lambert-Eaton myasthenic syndrome), HLA profiles are not the same.

ELIGIBILITY:
Inclusion Criteria:

* Presence of well-characterized antibodies in serum or cerebrospinal fluid;
* Clinical picture compatible with the detected antibody based on the literature;
* For PNS, cancer detected and compatible with the detected antibody based on the literature

Exclusion Criteria:

* Absence of complete clinicobiological data.
* Incongruences between antibody-clinics or antibody-cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years, having well-characterized anti-neural or anti-glial antibodies in serum and/or CSF detected in our laboratory, presenting with well-defined clinical pictures considered as associated with the aforementioned antibodies by a physician (neurologist) from the French Reference Center, including the presence of cancer in the case of paraneoplastic neurological syndromes; and whose clinical data is stocked at the database of our center.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Description of HLA alleles and haplotypes carrier frequencies in autoimmune encephalitis and paraneoplastic neurological syndromes. | 5 years. M1-M24: clinical database review, DNA extraction M25-M36: HLA analysis M37-M60: statistical analysis, combined analysis of genetic and clinical data
  Analyze the distribution of all HLA alleles at the level of the main HLA susceptibility loci, HLA A, B, C, DR, DQ and DP in all patients with AE or PNS.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Neurologique, Bron, France